CLINICAL TRIAL: NCT03861351
Title: A Multicenter, Non-controlled and Open-label Trial Following Subjects Implanted Bilaterally With the Toric Extended-depth-of-focus Mini WELL Toric Ready Intraocular Lens for 6 Months After the Second Eye Implant
Brief Title: Non-comparative Trial Following Participants Implanted Bilaterally With Mini WELL Toric Ready Intraocular Lens for 6 Months After the Second Eye Implant (FUSION)
Acronym: FUSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSM36
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Bilateral Cataract; Astigmatism
Keywords: Cataract; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Intervention Model Description: Men and women aged ≥ 18 years old suffering from bilateral cataract and astigmatism
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mini WELL Toric Ready intraocular lens (Experimental)
  Interventions: Device: Mini WELL Toric Ready intraocular lens

INTERVENTIONS:
Device: Mini WELL Toric Ready intraocular lens — The aim of cataract surgery is to remove the cloudy lens and replace it with the artificial intraocular lens called Mini WELL Toric Ready to correct presbyopia and to correct corneal astigmatism.

SUMMARY:
This is a multicenter, non-comparative trial following participants implanted bilaterally with the Mini WELL Toric Ready intraocular lens (IOL) for 6 months after the second eye implant.

The objective of the study is to evaluate the clinical performance of the Mini WELL Toric Ready intraocular lens (IOL), in particular, visual performance and rotational stability at 6 months following the second eye implantation in participants suffering from bilateral cataract with corneal astigmatism.

There are 2 hypotheses:

* Rotational Stability: the rotation of the Mini WELL Toric Ready IOL compared between Visit 0a (the day of surgery) and Visit 4 (120 180 days post-operative follow-up) shall be less than ±10° in 90% of the cases.
* Severe Visual Distortions: the rate of severe visual distortions for the Mini WELL Toric Ready IOL reported at 6 months postoperative will be less than 10 percents.

DETAILED DESCRIPTION:
This is an interventional, multicenter, non-comparative post-marketing clinical investigation in participants implanted bilaterally with the Mini WELL Toric Ready intraocular lens (IOL) for 6 months after the second eye implant.

The objective of this study is to evaluate the clinical performance of the Mini WELL Toric Ready IOL, in particular, visual performance and rotational stability at 6 months following second eye implantation.

The first hypothesis raised for this study is related to rotational stability. The rotation of the Mini WELL Toric Ready IOL compared between Visit 0a (the day of surgery) and Visit 4 (120 180 days post-operative follow-up) shall be less than ±10° in 90% of the cases.

The second hypothesis is regarding severe visual distortions. The rate of severe visual distortions for the Mini WELL Toric Ready IOL reported 6 months post-operative will be less than 10 percents.

The study will involve 45participants in 3 countries in order to achieve a target number of 38 evaluable participants completing the study.

This clinical study is composed of 9 scheduled visits. Following completion of the Informed Consent process, a pre-operative examination will take place to determine each patient's eligibility. Eligible patients, who wish to continue with the study, will be invited to undergo their first surgical procedure within 30 days. They will be required to undergo their second surgical procedure within 2 weeks of the initial operation. They will also be required to return for additional post-operative follow-up visits, 1-2 days after each eye surgery, 7-14 days after each eye surgery, 30-60 days after bilateral surgery and 120-180 days after bilateral surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older at the time of surgery and diagnosed with bilateral cataracts;
* Planned bilateral cataract removal by phacoemulsification;
* Preoperative total corneal astigmatism of 0.89 - 2.91 D, measured by corneal topography in both operative eyes;
* IOL power and cylinder requirement calculated by the specific web-based Mini Toric Calculator within the following range:
* Cylinder of: 1.50 D to 4.00 D
* Spherical Equivalent of: 18.00 to 28.00 D
* Willing and able to complete all required postoperative visits;
* Clear intraocular media other than cataract;
* Available for second-eye surgery within 2 weeks of the initial operation;
* Potential postoperative visual acuity of 0.3 logMAR in both eyes;
* Able to comprehend and sign a statement of informed consent consistent with local regulation for research in human subjects.

Exclusion Criteria:

* Irregular / asymmetric astigmatism;
* Significant irregular corneal aberration as demonstrated by corneal topography;
* Keratopathy / Kerectasia - any corneal abnormality, other than regular corneal astigmatism, including, but not limited to the following: keratoconus, keratoglobus, keratolysis, keratomalacia, keratomicosis and corneal plana;
* Any inflammation or edema (swelling) of the cornea, including but not limited to the following: keratitis, keratoconjuntivitis and keratouveitis;
* Subjects with diagnosed degenerative visual disorder (e.g. macular degeneration or other retinal disorders) that are predicted (by subjective assessment of the retina) to cause future acuity losses to a level worse than 0.3 logMAR;
* Subjects who may have reasonably been expected to require a secondary surgical intervention at any time during the study (other than Nd:YAG capsulotomy);
* Subjects in whom the intraocular lens might interfere with the ability to observe, diagnose or treat posterior segment conditions;
* Previous corneal refractive surgery;
* Other planned ocular surgery procedures, including, but not limited to LASIK, astigmatic keratotomy, retinal laser treatment and limbal relaxing incisions, for the duration of the study;
* Capsular or zonular abnormalities that may affect postoperative centration or tilt of the lens, including but not limited to the following: pseudo-exfoliation syndrome, chronic uveitis, Marfan's Syndrome;
* Absence of adequate capsular support for the implant of the intraocular lens in the capsular bag;
* Absence of adequate support for the lens from the posterior chamber or the zonule;
* Pupil abnormalities, including but not limited to the following: non-reactive, tonic pupils that do not dilatate under mesopic/scotopic conditions, abnormally shaped pupils or abnormally positioned pupils;
* Amblyopia;
* Clinically severe corneal dystrophy (e.g. epithelial, stromal, or endothelial dystrophy);
* Proliferative diabetic retinopathy;
* Microphthalmos;
* Suspected microbial infection;
* Previous retinal detachment;
* Previous corneal transplant;
* Optic nerve atrophy;
* Extremely shallow anterior chamber, not due to swollen cataract;
* Recurrent severe anterior or posterior segment inflammation of unknown aetiology (e.g. chronic uveitis);
* Iris neovascularization;
* Glaucoma (uncontrolled or controlled with medication);
* Aniridia or iris atrophy;
* Severe dry eye;
* Use of any systemic or topical drug known to interfere with visual performance;
* Subjects with any systemic disease that could increase operative risk or confound the outcomes (e.g. uncontrolled diabetes);
* Use of contact lens within the last 30 days before the preoperative visit;
* Vulnerable subjects (children <18 years, people in guardianship or trusteeship or inability to give an informed consent);
* Pregnant or lactating or planning a pregnancy at the time of enrolment;
* Subjects with psychiatric disorders that could confound the outcomes;
* Subjects participating in a concurrent clinical trial or if they have participated in an ophthalmology clinical trial within the last 30 days.

Intra-operative exclusion criteria:

* Irregularity and decentration of capsulorhexis;
* Other ocular surgery procedures, including, but not limited to LASIK, astigmatic keratotomy, retinal laser treatment and limbal relaxing incisions, for the duration of the study;
* Significant vitreous loss;
* Significant anterior chamber hyphema;
* Uncontrollable intraocular pressure (IOP);
* Zonular or capsular rupture;
* Ciliary sulcus, Bag-sulcus, sulcus-sulcus or unknown placement of the haptics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Intraocular lens (IOL) rotation | 6 months after second eye implant
  To evaluate the rotational stability of Mini WELL Toric Ready IOL.
Rate of severe visual distortions | 6 months after second eye implant
  To evaluate the visual performance of Mini WELL Toric Ready IOL.

OTHER OUTCOMES:
The rate of visual disturbances as detected with the Halometry test | 6 months after second eye implant
The rate of secondary surgical interventions (SSIs) related to the optical properties of the IOL for first and second operative eye separately | 6 months after second eye implant

CONTACTS AND LOCATIONS:
Locations (4):
- Service ophtalmologie Segment Antérieur- Hopital Pellegrin - CHU de Bordeaux, Bordeaux, France
- Universitäts-Augenklinik Heidelberg International Vision Correction Research Centre (IVCRC), Heidelberg, Germany
- Spain (2):
  - OFTALVIST CIO JEREZ Clínica Jerez (Cadiz), Jerez de la Frontera
  - Hospital Universitario Quirónsalud Madrid, Madrid